CLINICAL TRIAL: NCT06431698
Title: CORRECTION OF EAR DEFORMITIES IN NEWBORNS BY MODELING, COMPARISON OF TWO PROTOCOLS
Acronym: MOLDEAR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21-0023
Record Dates: First submitted 2024-05-22; First posted 2024-05-28 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-03

CONDITIONS: Ear Malformation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): Correction of deformation using the adjustable Earwell device
  Interventions: Device: adjustable Earwell device
- Intervention group (Experimental): Correction of deformation using the custom-made silicone device
  Interventions: Device: Custom-made silicone device

INTERVENTIONS:
Device: Custom-made silicone device — Correction of deformation using the custom-made silicone device
  Arms: Intervention group
Device: adjustable Earwell device — Correction of deformation using the adjustable Earwell device
  Arms: Control group

SUMMARY:
Evaluation of the non-inferiority of the custom-made device developed in the maxillofacial surgery department of Caen University Hospital compared to the device from the EarWell™ group

ELIGIBILITY:
Inclusion Criteria:

* Newborn, age between 8 days and 1 month
* newborn with ear malformation

Exclusion Criteria:

* Total chondrocutaneous agenesis of the ear
* polymalformative syndrome
* age greater than 4 weeks
* parental refusal

Max Age: 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 134 (Estimated)
Dates: Start 2023-07-31 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Subjective ear deformation score | baseline and 1 year after
  Evaluation of the non-inferiority of the custom-made device developed in the maxillofacial surgery department of Caen University Hospital compared to the device from the EarWell™ group.

CONTACTS AND LOCATIONS:
Locations (1):
- Caen University Hospital, Caen, N, France